CLINICAL TRIAL: NCT07110363
Title: An Open-label Phase Ib Study on the Safety, Tolerability, and Efficacy of BT02 in Treating Patients With Advanced Lung Cancer
Brief Title: A Clinical Study of BT02 in Treating Patients With Advanced Lung Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biotroy Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BT02-103
Record Dates: First submitted 2025-07-21; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Advanced Malignant Solid Tumor; Advanced Lung Cancer; Non-Small Cell Lung Cancer; Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- dose escalation and expansion (Experimental)
  Interventions: Drug: BT02

INTERVENTIONS:
Drug: BT02 — monoclonal antibody injection with intravenous administration every 2 or 3 weeks

SUMMARY:
The goal of this clinical trial is to assess whether an investigational treatment is safe and tolerable for patients with advanced lung cancer, and to get a preliminary idea of its effectiveness. Participants of all genders, aged between 18 and 75(inclusive), are eligible to join. These patients will receive the investigational drug intravenously every two weeks. If their condition doesn't worsen and they don't experience unbearable side effects, they can continue the treatment for up to two years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically confirmed locally advanced/unresectable or metastatic or recurrent non-small cell lung cancer (NSCLC, according to AJCC TNM staging) and advanced/unresectable limited-stage or extensive-stage small cell lung cancer (SCLC, according to VALG combined with AJCC TNM staging)，who have failed in the prior systemic therapy .
2. Adequate organ and hematologic function.
3. At least 1 extracranial measurable lesion.
4. An ECOG activity status score of 0-1.
5. A life expectancy of ≥ 3 months.
6. Eligible participants of childbearing potential (both males and females) must agree to using effective contraception throughout the study period.
7. Good compliance and willingness to follow up.

Exclusion Criteria:

1. Patients with sensitive mutations or gene fusions related to lung cancer.
2. Prior to the first dose , received systemic antitumor therapy, scheduled major surgical procedure within 4 weeks, received systemic immunostimulants within 5 half-lives and systemic corticosteroids or other immunosuppressive medications within 14 days.
3. A history of active autoimmune disease within the past 2 years.
4. A history of clinically significant cardiovascular disease, severe cardiac rhythm /conduction abnormalities or LVEF <50% . A history of severe pulmonary disease that may lead to severe episodes of dyspnea.
5. A severe acute or chronic infection when enrollment.
6. Remaining the toxic reaction in previous anti-tumor therapy that has not recovered to ≤ Grade 1 .
7. Unresolved > Grade 1 irAE or the history of a grade ≥ 3 irAE in previous immunotherapy, or known hypersensitivity to the formulation of the investigational product.
8. Clinically active CNS metastases or meningeal metastases.
9. A history of other type of malignancies.
10. Received a live attenuated vaccine within 28 days prior to the administration of the investigational product.
11. Poor compliance.
12. A history of alcohol or drugs abuse.
13. Current pregnancy or breastfeeding.
14. Other severe physical or mental illnesses or abnormal laboratory test results that the investigator deems unsuitable for participation in this study considering safety and compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Adverse events | through study completion, an average of 2 years
Dose limited toxicity incidence | Through the dose escalation phase , an average of 8 months
Maximum tolerated dose(MTD) | Through the dose escalation phase, an average of 8 months
Recommended Phase II dose (RP2D) | Through study completion, an average of 2 years

SECONDARY OUTCOMES:
Objective response rate (ORR) on tumor assessments | Through the study completion, an average of 2 years
Progression-free survival (PFS) on tumor assessments | Through the study completion，an average of 2 years
Overall survival (OS) on tumor assessments | Through the study completion, an average of 2 years
Duration of response (DoR) on tumor assessments | Through the study completion, an average of 2 years
Disease control rate (DCR) on tumor assessments | Through the study completion, an average of 2 years
Mean and median Area under the curve (AUC) of BT02 following first dose and repeated administration at each dose level | Through study completion, an average of 2 years
Mean and median Maximum concentration (Cmax) of BT02 following first dose and repeated administration at each dose level | Through study completion, an average of 2 years
ADA and NAb incidence | Through the study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, MD, Principal Investigator — Shanghai Chest Hospital of Shanghai Jiao Tong University

IPD SHARING:
Plan to Share IPD: Undecided